CLINICAL TRIAL: NCT00952055
Title: Effects of Standard Treatment of Acute Coronary Syndromes on Macrophage Activity as Measured by Serum Neopterin
Status: Terminated | Type: Observational
Why Stopped: 1) A delay in obtaining immunoassays to measure serum neopterin 2)altered relevance of the expected experimental results to clinical practice
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, Barbara George, Research Coordinator, Winthrop University Hospital
Other Study IDs: 03028
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Acute Coronary Syndrome
Keywords: neopterin; macrophage; inflammation
MeSH Terms: conditions — Acute Coronary Syndrome; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients diagnosed with acute coronary syndrome (ACS)

SUMMARY:
This is a prospective observational study focused on monitoring the effects of various treatment options for acute coronary syndrome (ACS) patients by measuring serum neopterin levels. Serum neopterin is a marker for measuring macrophage activation. Prior studies have illustrated that there are elevated serum neopterin levels in ACS. Patients enrolled are those with ACS. Blood samples are drawn at presentation, and at 72 hours after admission, or at office visits and at 72 hours later. Neopterin levels are measured via a commercially available assay..

DETAILED DESCRIPTION:
The study is a prospective observational study focused on monitoring the effects of various treatment options for acute coronary syndrome (ACS) patients by measuring serum neopterin levels. Serum neopterin is a marker for measuring macrophage activation. Prior studies have illustrated that there are elevated serum neopterin levels in ACS. The investigators' study focused on comparing different treatment arms with regard to their neopterin levels and correlating neopterin levels to the Thrombolysis in Myocardial Infarction (TIMI) risk score. Patients enrolled are those with ACS. Blood samples are drawn at presentation, and at 72 hours after admission, or at office visits and at 72 hours later. Neopterin levels are measured via a commercially available assay.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain and either ST segment elevation or depression > 0.1 mV in at least 2 contiguous electrocardiographic leads as well as elevation in troponin levels.

Exclusion Criteria:

* History of medical conditions known to alter neopterin concentrations in blood. The exclusion criteria includes:

  * renal failure,
  * history of HIV,
  * transplant patients,
  * active infections,
  * history of autoimmune disease,
  * malignancy,
  * phenylketonuria,
  * immune mediated liver disease, and
  * patients taking immunomodulating therapy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute cornary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 152 (Actual)
Dates: Start 2003-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Determine if serum neopterin is a useful marker in risk stratifying patients with acute coronary syndromes as it relates to vascular endothelial dysfunction. | 8 year study - 2011 anticipated study completion

SECONDARY OUTCOMES:
Evaluate whether serum neopterin is a useful marker in a similar manner as LPGD-S. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joshua DeLeon, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop-University Hospital, Mineola, New York, United States